CLINICAL TRIAL: NCT00758511
Title: Pain Reactivity to Non-pharmacological Interventions Across Repeated Routine Heel-Sticks in Preterm Infants in a Neonatal Intensive Care Unit
Acronym: PAMINA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University of Pittsburgh (Other); University Hospital, Zürich (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Eva Cignacco, PhD, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3200B1_122676; 3200B1_122676
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2010-02

CONDITIONS: Preterm Infants
Keywords: cortisol; pain; pain management; preterm infants; sucrose; facilitated tucking
MeSH Terms: conditions — Pain; Agnosia | interventions — Sucrose; Facilitated Tucking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Orally administrated 25%sucrose before,during and after heel stick across 5 heel sticks during the first 14 days of postnatal life
  Interventions: Procedure: 25% Sucrose
- 2 (Active Comparator): facilitated tucking before, during and after heel stick across 5 heel stick during the first 14 days of postnatal life
  Interventions: Procedure: facilitated tucking
- 3 (Active Comparator): orally administrated 25% sucrose AND facilitated tucking before, during and after heel stick across 5 heel sticks during the first 14 days of postnatal life
  Interventions: Procedure: Sucrose and facilitated tucking

INTERVENTIONS:
Procedure: 25% Sucrose — orally administrated 25%Sucrose before, during and after heel stick
  Arms: 1
Procedure: facilitated tucking — facilitated tucking before, during and after heel stick
  Arms: 2
Procedure: Sucrose and facilitated tucking — orally administrated 25%sucrose and facilitated tucking before, during and after heel stick
  Arms: 3

SUMMARY:
Switzerland is having one of the highest premature rates in Europa and most of the preterm neonates need neonatal intensive care. Up to 80% of the analgesic used in neonatal intensive care units are either "off label used" or "non-licensed" used. As an alternative approach non-pharmacological interventions for pain prevention and relief are increasingly being recommended for the prevention and treatment of mild and moderate pain in this population.

This multicenter pilot study will use a randomized three group,repeated measures design.

The primary aims of this study of premature neonates are to:

1.) Estimate effect sizes for the impact of the proposed interventions(facilitated tucking alone, sucrose alone and sucrose in combination with tucking)on pain reactivity.

2.) Examine the impact of gestational age on the estimates of efficacy 3.) Examine the impact of the numbers of painful procedures the infant experiences and the concurrent use of analgesic medications on the estimates of efficacy

DETAILED DESCRIPTION:
Background and significance:

Switzerland with its approximately 8% of premature births is having one of the highest premature rates in Europe and most of the preterm neonates need neonatal intensive care. Recur-rent neonatal pain and stress occur routinely during neonatal intensive care, particularly among the extremely low birth weight preterm neonates . It has become clear in recent years that the nervous system undergoes extensive development postnatally and there is increasing evidence that repeated exposure to pain, may lead to serious biobehavioral changes during the sensitive developmental phase of the central nervous system and that these changes may underlie long-term learning and behavior difficulties in this patient population. The frequency of exposure to pain and the adequate treatment of that pain are therefore important factors in later motor and cognitive development in preterm infants requiring intensive care. Pain treatment in infants is viewed as inadequate in the context of acute diagnostic and therapeutic procedures in the NICU. Up to 80% of the analgesic used in neonatal intensive care units (NICU) are either "off label used" or "non-licensed used". Secondary to significant side effects, associated with the use of analgesics drugs, health care providers are often reticence to administer these drugs in the NICU. As an alternative approach non-pharmacological interventions for pain prevention and relief are increasingly being recommended for the prevention and treatment of mild and moderate pain in this population. This type of intervention includes methods that involve reducing the sensitivity of the neonates during and after painful procedures, which have been shown to effectively reduce pain from minor procedures in neonates.

Although non-pharmacological interventions have been shown to be efficacious when tested during a single painful procedure there is a lack of evidence related to their efficacy after infants have being exposed to a high number of painful procedures and the accompanying chronic stress. To improve the clinical outcomes there is a critical need for accurate and efficient neonatal pain management for this highly vulnerable patient population.

Specific aims:

To determine the sample size needed for a larger randomized clinical trial (RCT) designed to compare the sustained impact of three non-pharmacological approaches on the pain reactivity of premature neo-nates in a NICU.

Design and methods:

This multicenter pilot study will use a randomized three group, repeated measures design. 72 premature infants from 24 0/7 to 32 0/7 weeks of gestation needing neonatal intensive care will be recruited during the first 2 days of life in three University Clinics (Bern, Basel, Zurich). The premature infants will be randomly assigned to one of three intervention groups (1) oral sucrose, (2) facilitated tucking, or (3) oral sucrose plus facilitated tucking. Sucrose is currently the standard of care in NICUs in Switzerland and will serve as the usual care control condition. The infants will be stratified into two gestational groups to examine the impact of gestational age on the effect size estimates. Five heel sticks across 12-14 days will be videotaped and pain will be rated by 4 independent raters, who are blinded to the data collection period. Raters will use the "Bernese Pain Scale for Neonates" to measure pain before, during and after the heel stick procedure. The physiologic data (heart rate and oxygen saturation) needed to complete the Bernese Pain Scale for Neonates will be down loaded from the clinical database for the same time frame as the neonate is videotaped. Near infrared spectroscopy (NIRS) will be performed during the painful procedures in the one site to measure differences in somatosensory cortical activation during heel sticks in infants managed with the three interventions at a baseline and across repeated heel sticks.

Expected value of the proposed project:

Adequate and efficient pain management is an important factor in later motor and cognitive development in preterm infants requiring intensive care. This pilot data will provide information about the sample size needed for a larger RCT. That study will compare the impact of the mentioned non-pharmacological interventions on pain reactivity across multiple painful procedures. In addition to examining their individual impact, we will evaluate the impact of using them in combination. The larger study will contribute to a better understanding of the efficacy of non-pharmacological pain relieving methods and their efficacy across repeated pain exposures. This pilot study is a collaborative effort of the disciplines of nursing science and neonatal medicine.

ELIGIBILITY:
Inclusion Criteria:

* must be born between 24 0/7 and 32 0/7 weeks of gestation
* must be hospitalized in the NICU
* it must be anticipated that they will need at least 5 routine heel sticks
* their parents give informed consent

Exclusion Criteria:

had a high-grade intraventricular hemorrhaging (grade III and IV);

* have a severe, life-threatening malformations;
* are suffering from any condition involving partial or total loss of sensitivity
* had a pHa < 7.00;
* had surgery for any reason; or
* have a congenital malformation affecting brain circulation or the cardiovascular system.

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pain reaction | first 14 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Eva EC Cignacco, PhD,MNSc, RM, Principal Investigator — Institute of Nursing Science, medical Faculty, University of Basel
Locations (1):
- Institute of Nursing Science Medical Faculty, University of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Gerull R, Cignacco E, Stoffel L, Sellam G, Nelle M. Physiological parameters after nonpharmacological analgesia in preterm infants: a randomized trial. Acta Paediatr. 2013 Aug;102(8):e368-73. doi: 10.1111/apa.12288. Epub 2013 May 28. PMID 23651076